CLINICAL TRIAL: NCT02124798
Title: An Open-Label Single-Arm Study to Evaluate the Reliability of an Autoinjector That Administers Belimumab Subcutaneously in Subjects With Systemic Lupus Erythematosus (SLE)
Brief Title: A Phase 2B Open-Label, Single-Arm, Repeat-Dose Study to Evaluate the Reliability of an Autoinjector
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 200339
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Subcutaneous; Autoinjector; Belimumab; Real-Life Use Study; Reliability
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Subjects will self-administer belimumab SC into thigh or abdomen using the autoinjector device for 8 weekly doses; 4 of the doses will be administered under observation in the clinic and 4 of the doses will be administered outside the clinic and without observation
  Interventions: Device: Belimumab autoinjector

INTERVENTIONS:
Device: Belimumab autoinjector — Single use, disposable autoinjector assembled with the prefilled syringe containing the drug product belimumab with unit dose strength of 200mg/mL and 1 mL will be given as a once weekly SC dose

SUMMARY:
The primary objective of this study is to assess the suitability of the autoinjector for self-administration of belimumab by subjects with SLE in real-life conditions. The study will assess the use of the autoinjector inside the clinic setting and outside the clinic setting. The study will also assess the safety and tolerability of belimumab administered subcutaneously (SC) via the autoinjector. Subjects will self-administer belimumab SC into the thigh or abdomen using the autoinjector device for 8 weekly doses. Subjects will return for a follow-up visit 4 weeks after the last SC dose of belimumab. All injections will be assessed by the investigators for success based on direct observation and/or the subject diary. A total of 118 subjects (treated with at least one dose of study drug) are planned to be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged at least 18 years at the time of signing the informed consent.
* Have a clinical diagnosis of SLE according to the American College of Rheumatology (ACR) criteria.
* Active, autoantibody positive SLE, defined as the presence of anti nuclear antibody (ANA) or anti-double strand deoxyribonucleic acid (dsDNA) antibodies (at screening or historically).
* Are on a SLE treatment regimen including intravenous (IV) belimumab every 28 days for at least three 28-day cycles. Day 0 (i.e., day of first dose of study agent) should be scheduled about 2 weeks after the last dose IV dose of belimumab but may be scheduled 1 week and up to 4 weeks after the last IV dose.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy (for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records); or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] >40 milli international unit/milliliter [MIU/mL] and estradiol <40 picogram/mL [<147 picomoles/Liter] is confirmatory). (Females on hormone replacement therapy [HRT] and whose menopausal status is in doubt will be required to use one of the contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2 4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.); Child-bearing potential with negative pregnancy test as determined by serum human chorionic gonadotropin (hCG) test at screening and urine hCG test prior to dosing; Agrees to use one of the contraception methods for 2 weeks prior to the day of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until Day 112; OR has only same-sex partners, when this is her preferred and usual lifestyle
* Alanine aminotransferase (ALT) <2x upper limit of normal (ULN), alkaline phosphatase and bilirubin <=1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Have previously participated in a study of SC belimumab.
* Have received a live vaccine within 30 days of Day 0 or anticipate receipt of a live vaccine during the study or within 120 days after the last injection of study drug.
* Have received a non-biologic investigational agent within 60 days of Day 0.
* Have severe active central nervous system (CNS) lupus (including seizures, psychosis, organic brain syndrome, cerebrovascular accident (CVA), cerebritis or CNS vasculitis requiring therapeutic intervention within 60 days of Day 0.
* Have clinical evidence of significant unstable or uncontrolled acute or chronic diseases not due to SLE (i.e., cardiovascular, pulmonary, hematologic, gastrointestinal, hepatic, renal, neurological, malignancy, or infectious diseases) which, in the opinion of the principal investigator, could confound the results of the study or put the subject at undue risk.
* Have a planned surgical procedure
* History of any other medical disease (e.g., cardiopulmonary), laboratory abnormality, that, in the opinion of the investigator, makes the subject unsuitable for the study.
* Have required management of acute or chronic infections, as follows: Currently on any suppressive therapy for a chronic infection (such as tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster, and atypical mycobacteria); Hospitalization for treatment of infection within 60 days of Day 0; Use of parenteral (IV or intramascular [IM]) antibiotics (antibacterials, antivirals, anti-fungals, or anti-parasitic agents) within 60 days of Day 0.
* History of or a positive test for human immuno virus (HIV) at Screening.
* A positive Hepatitis B surface antigen or Hepatitis B core antibody, or positive Hepatitis C antibody result within 3 months of Screening or positive at Screening.
* Have an Immunoglobulin A (IgA) deficiency (IgA level <10 milligrams/deciliter).
* Have a Grade 3 or greater laboratory abnormality based on the Adverse Event Severity Grading except for the following that are allowed: Stable Grade 3 prothrombin time (PT) secondary to warfarin treatment; Stable Grade 3 partial thromboplastin time (PTT) due to lupus anticoagulant and not related to liver disease or anti-coagulant therapy; Stable Grade 3/4 proteinuria (<=6 grams/24 hour equivalent by spot urine protein to creatinine ratio allowed); Stable Grade 3 hypoalbuminemia due to lupus nephritis, and not related to liver disease or malnutrition; Stable Grade 3 gamma glutamyl transferase (GGT) elevation due to lupus hepatitis, and not related to alcoholic liver disease, uncontrolled diabetes, or viral hepatitis. If present, any abnormalities in the ALT and/or aspartate aminotransferase (AST) must be<= Grade 2; Stable Grade 3 neutropenia or stable Grade 3 white blood cell count. Note: All Grade 3 or greater laboratory abnormalities will be flagged in the laboratory report. Therefore the above exceptions will be determined by the Investigator and Medical Monitor.
* Have a history of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins, or monoclonal antibodies
* Have evidence of serious suicide risk including any history of suicidal behavior in the last 6 months, or who in the investigator's opinion, pose a significant suicide risk
* Have current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within 364 days prior to Day 0
* Are unable to administer study agent by SC injection.
* In the opinion of the investigator, any subject who is unable to read and/or would not be able to complete a patient diary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2014-05-20 (Actual); Primary Completion 2015-04-13 (Actual); Study Completion 2015-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (25):
- United States (25):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Tuscaloosa, Alabama
  - GSK Investigational Site, Gilbert, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, San Leandro, California
  - GSK Investigational Site, Tustin, California
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Lansing, Michigan
  - GSK Investigational Site, Flowood, Mississippi
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Smithtown, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Duncansville, Pennsylvania
  - GSK Investigational Site, Wyomissing, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Webster, Texas
  - GSK Investigational Site, Beckley, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 200339 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200339 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 200339 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200339 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 200339 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200339 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200339 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a study in participants with Systemic Lupus Erythematosus (SLE). The study was conducted at 27 centers in the United States from 20 May 2014 to 13 April 2015.
Pre-assignment Details: A total of 119 participants were screened out of which only 95 were enrolled to the study treatment. 25 were screen failures the reasons for which were did not meet inclusion/exclusion criteria (23), lost to follow up (1), withdrew consent (1).
Groups:
- Total: Eligible participants self administered once weekly dose of 200 milligram per milliliter (mg/mL), of belimumab subcutaneously (SC) into thigh or abdomen with an auto-injector device for 8 weeks. Of which 4 of the doses were administered under observation in the clinic (week 1, 2, 4 and week 8) under the supervision of investigator and 4 of the doses were administered outside the clinic and without observation (week 3, 5,6 and week 7).
Period: Overall Study
Arm/Group | Total
Started | 95
Completed | 91
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Belimumab 200mg Auto Injector: Eligible participants self administered once weekly dose of 200 mg/mL, of belimumab SC into thigh or abdomen with an auto-injector device for 8 weeks. Of which 4 of the doses were administered under observation in the clinic (week 1, 2, 4 and week 8) under the supervision of investigator and 4 of the doses were administered outside the clinic and without observation (week 3, 5,6 and week 7).
Arm/Group | Belimumab 200mg Auto Injector
Number analyzed (Participants) | 95
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.8 (12.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 69
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Successfully Able to Self-administer Their Observed First and Second Doses in Weeks 1 and 2 (Inside Clinic)
Description: The primary objective was to assess the suitability of the auto injector for self-administration of belimumab. An overall assessment of usability and reliability for the device was determined by assessing the rate of successfully complete self-administered injections relative to attempted ones. The assessment for the parameter, drug successfully injected was elicited by a Yes/No response. The participants who were able to administer injections inside and outside of the clinic without assistance were included.
Time Frame: Weeks 1 and 2 (Inside clinic)
Population: The intention-to-treat (ITT) population was defined as all participants who were enrolled and treated with at least 1 dose of belimumab. Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Belimumab 200mg Auto Injector
Number analyzed (Participants) | 90
Participants
  Week 1 and 2, YES | 89
  Week 1 and 2, NO | 1

2. Secondary Outcome: Number of Participants Successfully Able to Self-administer Their Observed Doses in Weeks 4 and 8 (Inside Clinic)
Description: The main objective was to assess the suitability of the auto injector for self-administration of belimumab by participants with SLE. An overall assessment of usability and reliability for the device was determined by assessing the rate of successfully complete self-administered injections relative to attempted ones. The assessment for the parameter, drug successfully injected was elicited by a Yes/No response. The participants who were able to administer injections inside and outside of the clinic without assistance were included.
Time Frame: Weeks 4 and 8 (Inside clinic)
Population: ITT population. Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Belimumab 200mg Auto Injector
Number analyzed (Participants) | 87
Participants
  Week 4 and 8, YES | 85
  Week 4 and 8, NO | 2

3. Secondary Outcome: Number of Participants Who Reported They Were Successfully Able to Self-administer Their Doses Outside the Clinic Setting in Weeks 3, 5, 6, and 7 (Outside Clinic)
Description: Assessment was performed for suitability of the auto injector for self-administration of belimumab by participant with SLE outside the clinic setting. An overall assessment of usability and reliability for the device was determined by assessing the rate of successfully complete self-administered injections relative to attempted ones. The assessment for the parameter, drug successfully injected was elicited by a Yes/No response. The participants who were able to administer injections outside of the clinic without assistance were included.
Time Frame: Weeks 3, 5, 6, and 7 (Outside clinic)
Population: ITT population. Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Belimumab 200mg Auto Injector
Number analyzed (Participants) | 87
Participants
  Weeks 3, 5, 6 and 7, YES | 81
  Weeks 3, 5, 6 and 7, NO | 6

ADVERSE EVENTS:
Time Frame: From start of treatment (Day 0, week 1) up to week 12
Description: All adverse events (AEs) and serious AEs (SAEs) were collected from the first dosing day (Day 0) to Week 12. The ITT population was used for analysis.
Arm/Group | Belimumab 200mg Auto Injector
All-Cause Mortality (participants affected / at risk) | 0/95
Serious Adverse Events (participants affected / at risk) | 4/95
Other Adverse Events (participants affected / at risk) | 28/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belimumab 200mg Auto Injector (N=95)
Anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Pneumonia (Infections and infestations) | 1
Postoperative abscess (Infections and infestations) | 1
Pyrexia (General disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Belimumab 200mg Auto Injector (N=95)
Bronchitis (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 3
Gastroenteritis viral (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Nausea (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 2
Fatigue (General disorders) | 2
Injection site erythema (General disorders) | 2
Malaise (General disorders) | 2
Headache (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.